CLINICAL TRIAL: NCT00470080
Title: Randomised Trial of Eutectic Mixture of Local Anaesthetics Cream and Oral Sucrose Solution for Venepuncture in Preterm Infants
Brief Title: Randomised Trial of Eutectic Mixture of Local Anaesthetics Cream and Oral Sucrose Solution for Venepuncture
Acronym: VIEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick VACHER, Department Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P060501
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2007-05

CONDITIONS: Pain
Keywords: Venepuncture; Pain; Emla cream; Oral sucrose solution; Premature infant; Premature infant admitted to the care baby unit were; included in the study.; Programed venepuncture is performed with analgesia.
MeSH Terms: conditions — Pain; Premature Birth | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): venepuncture
  Interventions: Procedure: venepuncture

INTERVENTIONS:
Procedure: venepuncture — venepuncture

SUMMARY:
This randomized bicentric trial will investigate the efficacy of topical EMLA cream with oral sucrose solution compared to oral sucrose solution alone before venepuncture in preterm infants.

DETAILED DESCRIPTION:
Venepuncture is a painful procedure commonly performed in premature infants. Nonpharmacological intervention (oral sucrose solution) can reduce neonatal pain. EMLA cream is an oil in water emulsion of an eutectic mixture of prilocaine and lignocaine; it is an local anesthetic cream. Very few reports have looked at the efficacy of EMLA in preterm infants.

This randomized bicentric trial will investigate the efficacy of topical EMLA cream with oral sucrose solution compared to oral sucrose solution alone before venepuncture in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants (gestational age between 26 and 37 weeks)
* programmed venepuncture
* APGAR score (M5)≥ 7
* enteral feeding
* written parental consent

Exclusion Criteria:

* infant requiring oxygen
* analgesia or sedation or drugs causing methaemoglobinaemia
* congenital porphyria
* G6PD deficit
* multi organ failure
* convulsion
* dermatosis

Ages: 26 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2007-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Association of oral sucrose solution and EMLA cream will reduce pain responses in premature infant for venepuncture.A combination of physiological and behavioural responses are used for the measurement of pain in neonates : DAN score and PIPP. | in 24 hours
  Association of oral sucrose solution and EMLA cream will reduce pain responses in premature infant for venepuncture.A combination of physiological and behavioural responses are used for the measurement of pain in neonates : DAN score and PIPP.

SECONDARY OUTCOMES:
Clinical units providing health care in newborns develop written guidelines and protocols for the management of neonatal pain, like venepuncture with the combination of sucrose oral solution and EMLA cream. | in the 24 hours
  Clinical units providing health care in newborns develop written guidelines and protocols for the management of neonatal pain, like venepuncture with the combination of sucrose oral solution and EMLA cream.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BIRAN, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CHU Armand Trousseau, Paris, France

REFERENCES:
- [Result] Acharya AB, Annamali S, Taub NA, Field D. Oral sucrose analgesia for preterm infant venepuncture. Arch Dis Child Fetal Neonatal Ed. 2004 Jan;89(1):F17-8. doi: 10.1136/fn.89.1.f17. No abstract available. PMID 14711847
- [Result] Acharya AB, Bustani PC, Phillips JD, Taub NA, Beattie RM. Randomised controlled trial of eutectic mixture of local anaesthetics cream for venepuncture in healthy preterm infants. Arch Dis Child Fetal Neonatal Ed. 1998 Mar;78(2):F138-42. doi: 10.1136/fn.78.2.f138. PMID 9577286